CLINICAL TRIAL: NCT02229084
Title: A Combined Phase I/II Feasibility-and-Efficacy Study of a Carbohydrate Mimotope-based Vaccine With MONTANIDE™ ISA 51 VG Combined With Neoadjuvant Chemotherapy
Brief Title: Vaccination of High Risk Breast Cancer Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202556
Record Dates: First submitted 2014-08-26; First posted 2014-08-29 (Estimated); Results first posted 2024-05-23 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer; Breast Neoplasms
Keywords: clinical stage I, II or III; ER postive; HER2 negative
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Cyclophosphamide; Docetaxel

STUDY DESIGN:
Intervention Model Description: This combined Phase I/II feasibility-and-efficacy study will have three parts. Part 1 will be a Phase I evaluation of the safety, tolerability, and feasibility of the Chemovax to assess the timing of vaccination relative to chemotherapy. Five different Chemovax schedules (Schedule A, B, C, D, and E) will be sequentially evaluated. Once such a feasible schedule is identified, the study will proceed with its second and third parts. Part 2 (primary efficacy) and Part 3 (expanded efficacy) will respectively constitute Stages 1 and 2 of the Phase II primary-efficacy evaluation of Chemovax using a Simon optimal two-stage design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part 1 - Chemovax Schedule A (Experimental): Feasibility - Chemovax schedule A: Subjects will receive the first cycle of chemotherapy along with the first injection of P10s-PADRE/MONTANIDE™ ISA 51 VG vaccine on week 1, the subsequent two injections of the vaccine one week apart (week 2 and 3), second cycle of chemotherapy on week 4, and subsequent cycles of chemotherapy every 21 days (week 7,10,13,16,19,22).
  Interventions: Biological: P10s-PADRE/ MONTANIDE™ ISA 51 VG; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Docetaxel
- Part 1 - Chemovax Schedule B (Experimental): Feasibility - Chemovax Schedule B: Subjects will receive the first cycle of chemotherapy on week 1, the first injection of P10s-PADRE/MONTANIDE™ ISA 51 VG vaccine on week 2, the subsequent two injections of the vaccine one week apart (week 3 and 4), second cycle of chemotherapy on week 4 (along with second vaccine injection) and subsequent cycles of chemotherapy every 21 days (week 7,10,13,16,19,22).
  Interventions: Biological: P10s-PADRE/ MONTANIDE™ ISA 51 VG; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Docetaxel
- Part 1 - Chemovax Schedule C (Experimental): Feasibility - Chemovax Schedule C: Subjects will receive three weekly injections of P10s-PADRE/MONTANIDE™ ISA 51 VG vaccine (week 1,2,3), then first cycle of chemotherapy (week 4), and subsequent cycles of chemotherapy every 21 days (week 7,10,13,16,19,22,25).
  Interventions: Biological: P10s-PADRE/ MONTANIDE™ ISA 51 VG; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Docetaxel
- Part 1 - Chemovax Schedule D (Experimental): Feasibility - Chemovax Schedule D: Subjects will receive the first injection of vaccine on week 1, the subsequent two injections of the P10s-PADRE/MONTANIDE™ ISA 51 VG vaccine one week apart (week 2 and 3), the first cycle of chemotherapy on week 2 (along with second vaccine injection) and subsequent cycles of chemotherapy every 21 days (week 5,8,11,14,17,20,23).
  Interventions: Biological: P10s-PADRE/ MONTANIDE™ ISA 51 VG; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Docetaxel
- Part 1 - Chemovax Schedule E (Experimental): Feasibility - Chemovax Schedule E: Subjects will receive the first injection of vaccine on week 1, the subsequent two injections of the P10s-PADRE/MONTANIDE™ ISA 51 VG vaccine one week apart (week 2 and 3), the first cycle of chemotherapy on week 3 (along with third vaccine injection) and subsequent cycles of chemotherapy every 21 days (week 6,9,12,15,18,21,24).
  Interventions: Biological: P10s-PADRE/ MONTANIDE™ ISA 51 VG; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Docetaxel
- Part 2 - Chemovax Schedule C (Experimental): Primary Efficacy - Chemovax Schedule C: Subjects will receive three weekly injections of P10s-PADRE/MONTANIDE™ ISA 51 VG vaccine (week 1,2,3), then first cycle of chemotherapy (week 4), and subsequent cycles of chemotherapy every 21 days (week 7,10,13,16,19,22,25).
  Interventions: Biological: P10s-PADRE/ MONTANIDE™ ISA 51 VG; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Docetaxel
- Part 3 - Chemovax Schedule C (Experimental): Expanded Efficacy - Chemovax Schedule C: Subjects will receive three weekly injections of P10s-PADRE/MONTANIDE™ ISA 51 VG vaccine (week 1,2,3), then first cycle of chemotherapy (week 4), and subsequent cycles of chemotherapy every 21 days (week 7,10,13,16,19,22,25).
  Interventions: Biological: P10s-PADRE/ MONTANIDE™ ISA 51 VG; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Docetaxel

INTERVENTIONS:
Biological: P10s-PADRE/ MONTANIDE™ ISA 51 VG — Eligible subjects will be enrolled and immunized by SC administration of P10s-PADRE vaccine on each of 3 separate occasions concurrent with chemotherapy.
Drug: Doxorubicin — Doxorubicin (60 mg/m2) and cyclophosphamide (600 mg/m2) (AC) will be administered concurrently every three weeks for four cycles followed by docetaxel (75 mg/m2) every three weeks for four cycles.
Drug: Cyclophosphamide — Doxorubicin (60 mg/m2) and cyclophosphamide (600 mg/m2) (AC) will be administered concurrently every three weeks for four cycles followed by docetaxel (75 mg/m2) every three weeks for four cycles.
Drug: Docetaxel — Doxorubicin (60 mg/m2) and cyclophosphamide (600 mg/m2) (AC) will be administered concurrently every three weeks for four cycles followed by docetaxel (75 mg/m2) every three weeks for four cycles.
  If docetaxel is not tolerated, paclitaxel (175mg/m2) may be used in its place.

SUMMARY:
The purpose of this study is to evaluate a new investigational cancer vaccine, P10s-PADRE in combination with standard neoadjuvant chemotherapy and surgery in patients with clinical stage I, II or III estrogen-receptor (ER)-positive, HER2-negative breast cancer.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate an investigational agent, P10s-PADRE, a peptide mimotope-based vaccine, in combination with standard neoadjuvant chemotherapy in patients with clinical stage I, II or III estrogen-receptor (ER)-positive, HER2-negative breast cancer.

This is a single-arm, multi-site Phase I/II study designed with the two goals being (1) to evaluate the feasibility of combining vaccination with the P10s-PADRE formulation with neoadjuvant chemotherapy and (2) to determine if the polymerase chain reaction (pCR) rate among ER-positive, HER2-negativebreast-cancer patients treated with the combination is significantly higher than the 8% rate observed among ER-positive breast-cancer subjects in a pooled analysis of seven randomized clinical trials. P10s-PADRE vaccine with MONTANIDE™ ISA 51 VG as adjuvant will be given in combination with neoadjuvant chemotherapy in female patients with clinical stage I, II or III ER-positive, HER2-negative breast cancer.

This combined Phase I/II feasibility-and-efficacy study will have three parts. Its first part will be a Phase I evaluation of the safety, tolerability, and feasibility of eliciting adequate IgG response with P10s-PADRE when administered in combination with SoC neoadjuvant chemotherapy. The study's second and third parts will respectively constitute Stages 1 and 2 of the Phase II primary-efficacy evaluation of Chemovax using a Simon optimal two-stage design

To evaluate the feasibility of eliciting adequate immune response with P10s-PADRE when it is administered in combination with neoadjuvant chemotherapy, we will sequentially evaluate different schedules of vaccination relative to chemotherapy, and stop evaluating as soon as we have identified a feasible schedule. To this end, we have defined five different Chemovax schedules, and named them A, B, C, D, and E;

ELIGIBILITY:
Inclusion Criteria:

* Females of all races with clinical stage I, II, or III ER-positive, HER2 negative breast cancer who will undergo SoC neoadjuvant treatment.
* Age 18 years and older.
* ECOG Performance Status 0 or 1.
* White blood cell (WBC) count ≥ 3,000/mm3 within 3 weeks prior to registration.
* Platelet count ≥ 100,000/mm3 within 3 weeks prior to registration.
* Bilirubin ≤ 2 x institutional upper limit (IUL) of normal obtained within 3 weeks prior to registration.
* Serum glutamic-oxaloacetic transaminase (SGOT) or aspartate aminotransferase test (AST) ≤ 2 x IUL of normal obtained within 3 weeks prior to registration.
* Serum glutamic-pyruvic transaminase (SGPT) or alanine aminotransferase test (ALT) ≤ 2 x IUL of normal obtained within 3 weeks prior to registration.
* Serum creatinine ≤ 1.8 mg/dL obtained within 3 weeks prior to registration.
* Must sign an informed consent document approved by the UAMS IRB.

Exclusion Criteria:

* ER-negative, HER2-positive, inflammatory, metastatic, stage IV or recurrent breast cancer
* Active infection requiring treatment with antibiotics.
* Existing diagnosis or history of organic brain syndrome that might preclude participation in the full protocol.
* Existing diagnosis or history of significant impairment of basal cognitive function that might preclude participation in the full protocol.
* Other current malignancies. Subjects with prior history at any time of any in situ cancer, including lobular carcinoma of the breast in situ, cervical cancer in situ, atypical melanocytic hyperplasia or Clark I melanoma in situ or basal or squamous skin cancer are eligible, provided they are disease-free at the time of registration. Subjects with other malignancies are eligible if they have been continuously disease free for ≥ 5 years prior to the time of registration.
* Active autoimmune disorders or conditions of immunosuppression; Existing diagnosis or history of autoimmune disorders or conditions of immunosuppression that have been in remission for less than 6 months
* Treatment with corticosteroids, including oral steroids (i.e. prednisone, dexamethasone [except when used as an antiemetic in SoC therapy]), continuous use of topical steroid creams or ointments or any steroid-containing inhalers. Subjects who discontinue the use of these classes of medication for at least 6 weeks prior to registration are eligible if, in the judgment of the treating physician, the subject is not likely to require these classes of drugs during the treatment period. Replacement doses of steroids for subjects with adrenal insufficiency are allowed.
* Pregnancy or breastfeeding (due to the unknown effects of peptide/mimotope vaccines on a fetus or infant). Women of childbearing potential must have a negative urine pregnancy test within 72 hours prior to starting week 1 and must be counseled to use an accepted and effective method of contraception (including abstinence) while on treatment and for a period of 18 months after completing or discontinuing treatment. Accepted methods of contraception include tubal ligation, oral contraceptives, barrier methods, IUDs, and abstinence.
* Any other significant medical or psychiatric conditions, which, in the opinion of the enrolling investigator, may interfere with consent or compliance of the treatment regimen.
* Enrollment in any other clinical trial using investigational drug products or devices prior to first post-surgery study lab. Concurrent enrollment in observational studies is allowed.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2015-01-14 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sri Obulareddy, MD, Principal Investigator — University of Arkansas
Locations (2):
- United States (2):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas

REFERENCES:
- [Derived] Hernandez Puente CV, Hsu PC, Rogers LJ, Jousheghany F, Siegel E, Kadlubar SA, Beck JT, Makhoul I, Hutchins LF, Kieber-Emmons T, Monzavi-Karbassi B. Association of DNA-Methylation Profiles With Immune Responses Elicited in Breast Cancer Patients Immunized With a Carbohydrate-Mimicking Peptide: A Pilot Study. Front Oncol. 2020 Jun 5;10:879. doi: 10.3389/fonc.2020.00879. eCollection 2020. PMID 32582547

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential subjects were recruited from the Winthrop P Rockefeller Cancer Institute on the University of Arkansas for Medical Sciences campus and clinics at Highlands Oncology Group.
Groups:
- Part 1 - Chemovax Schedule A: Feasibility - Chemovax schedule A: Subjects will receive the first cycle of chemotherapy along with the first injection of P10s-PADRE/MONTANIDE™ ISA 51 VG vaccine on week 1, the subsequent two injections of the vaccine one week apart (week 2 and 3), second cycle of chemotherapy on week 4, and subsequent cycles of chemotherapy every 21 days (week 7,10,13,16,19,22).
  Chemovax - P10s-PADRE/ MONTANIDE™ ISA 51 VG + Doxorubicin + Cyclophosphamide + Docetaxel (or Paclitaxel): Eligible subjects will be enrolled and immunized by SC administration of P10s-PADRE vaccine on each of 3 separate occasions over a three-week period.
- Part 1 - Chemovax Schedule B: Feasibility - Chemovax Schedule B: Subjects will receive the first cycle of chemotherapy on week 1, the first injection of P10s-PADRE/MONTANIDE™ ISA 51 VG vaccine on week 2, the subsequent two injections of the vaccine one week apart (week 3 and 4), second cycle of chemotherapy on week 4 (along with second vaccine injection) and subsequent cycles of chemotherapy every 21 days (week 7,10,13,16,19,22).
  Chemovax - P10s-PADRE/ MONTANIDE™ ISA 51 VG + Doxorubicin + Cyclophosphamide + Docetaxel (or Paclitaxel): Eligible subjects will be enrolled and immunized by SC administration of P10s-PADRE vaccine on each of 3 separate occasions over a three-week period.
- Part 1 - Chemovax Schedule C: Feasibility - Chemovax Schedule C: Subjects will receive three weekly injections of P10s-PADRE/MONTANIDE™ ISA 51 VG vaccine (week 1,2,3), then first cycle of chemotherapy (week 4), and subsequent cycles of chemotherapy every 21 days (week 7,10,13,16,19,22,25).
  Chemovax - P10s-PADRE/ MONTANIDE™ ISA 51 VG + Doxorubicin + Cyclophosphamide + Docetaxel (or Paclitaxel): Eligible subjects will be enrolled and immunized by SC administration of P10s-PADRE vaccine on each of 3 separate occasions over a three-week period.
- Part 1 - Chemovax Schedule D: Feasibility - Chemovax Schedule D: Subjects will receive the first injection of vaccine on week 1, the subsequent two injections of the P10s-PADRE/MONTANIDE™ ISA 51 VG vaccine one week apart (week 2 and 3), the first cycle of chemotherapy on week 2 (along with second vaccine injection) and subsequent cycles of chemotherapy every 21 days (week 5,8,11,14,17,20,23).
  Chemovax - P10s-PADRE/ MONTANIDE™ ISA 51 VG + Doxorubicin + Cyclophosphamide + Docetaxel (or Paclitaxel): Eligible subjects will be enrolled and immunized by SC administration of P10s-PADRE vaccine on each of 3 separate occasions over a three-week period.
- Part 1 - Chemovax Schedule E: Feasibility - Chemovax Schedule E: Subjects will receive the first injection of vaccine on week 1, the subsequent two injections of the P10s-PADRE/MONTANIDE™ ISA 51 VG vaccine one week apart (week 2 and 3), the first cycle of chemotherapy on week 3 (along with third vaccine injection) and subsequent cycles of chemotherapy every 21 days (week 6,9,12,15,18,21,24).
  Chemovax - P10s-PADRE/ MONTANIDE™ ISA 51 VG + Doxorubicin + Cyclophosphamide + Docetaxel (or Paclitaxel): Eligible subjects will be enrolled and immunized by SC administration of P10s-PADRE vaccine on each of 3 separate occasions over a three-week period.
- Part 2 - Chemovax Schedule C: Primary Efficacy - Chemovax Schedule C: Subjects will receive three weekly injections of P10s-PADRE/MONTANIDE™ ISA 51 VG vaccine (week 1,2,3), then first cycle of chemotherapy (week 4), and subsequent cycles of chemotherapy every 21 days (week 7,10,13,16,19,22,25).
  Chemovax - P10s-PADRE/ MONTANIDE™ ISA 51 VG + Doxorubicin + Cyclophosphamide + Docetaxel (or Paclitaxel): Eligible subjects will be enrolled and immunized by SC administration of P10s-PADRE vaccine on each of 3 separate occasions over a three-week period.
- Part 3 - Chemovax Schedule C: Expanded Efficacy - Chemovax Schedule C: Subjects will receive three weekly injections of P10s-PADRE/MONTANIDE™ ISA 51 VG vaccine (week 1,2,3), then first cycle of chemotherapy (week 4), and subsequent cycles of chemotherapy every 21 days (week 7,10,13,16,19,22,25
  Chemovax - P10s-PADRE/ MONTANIDE™ ISA 51 VG + Doxorubicin + Cyclophosphamide + Docetaxel (or Paclitaxel): Eligible subjects will be enrolled and immunized by SC administration of P10s-PADRE vaccine on each of 3 separate occasions over a three-week period.
Period: Overall Study
Arm/Group | Part 1 - Chemovax Schedule A | Part 1 - Chemovax Schedule B | Part 1 - Chemovax Schedule C | Part 1 - Chemovax Schedule D | Part 1 - Chemovax Schedule E | Part 2 - Chemovax Schedule C | Part 3 - Chemovax Schedule C
Started | 5 | 5 | 5 | 5 | 5 | 19 | 14
Completed | 4 | 5 | 3 | 3 | 1 | 18 | 10
Not Completed | 1 | 0 | 2 | 2 | 4 | 1 | 4
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 3 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 1 | 1 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Part 3 - Chemovax Schedule C: Expanded Efficacy - Chemovax Schedule C: Subjects will receive three weekly injections of P10s-PADRE/MONTANIDE™ ISA 51 VG vaccine (week 1,2,3), then first cycle of chemotherapy (week 4), and subsequent cycles of chemotherapy every 21 days (week 7,10,13,16,19,22,25)..
  Chemovax - P10s-PADRE/ MONTANIDE™ ISA 51 VG + Doxorubicin + Cyclophosphamide + Docetaxel (or Paclitaxel): Eligible subjects will be enrolled and immunized by SC administration of P10s-PADRE vaccine on each of 3 separate occasions over a three-week period.
- Total: Total of all reporting groups
Arm/Group | Part 1 - Chemovax Schedule A | Part 1 - Chemovax Schedule B | Part 1 - Chemovax Schedule C | Part 1 - Chemovax Schedule D | Part 1 - Chemovax Schedule E | Part 2 - Chemovax Schedule C | Part 3 - Chemovax Schedule C | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 19 | 14 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 4 | 3 | 4 | 17 | 13 | 49
  >=65 years | 1 | 1 | 1 | 2 | 1 | 2 | 1 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (12.37) | 53 (10.2) | 57.6 (11.69) | 54.8 (15.42) | 43.4 (15.24) | 52.58 (10.73) | 46.86 (10.73) | 50.15 (10.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 5 | 5 | 5 | 19 | 14 | 58
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 10 | 6 | 16
  Unknown or Not Reported | 5 | 5 | 5 | 5 | 5 | 9 | 6 | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
  Native Hawaiian or Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 0 | 5 | 3 | 9
  White | 5 | 3 | 5 | 5 | 5 | 14 | 8 | 45
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Central Arkansas at University of Arkansas for Medical Sciences | 5 | 5 | 2 | 1 | 0 | 10 | 14 | 37
  United States: Northwest Arkansas at Highlands Oncology Group | 0 | 0 | 3 | 4 | 5 | 9 | 0 | 21
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Measure of how cancer affects a person's day-to-day life (https://ecog-acrin.org/resources/ecog-performance-status/). In this study, having a score of 0-1 was a criterion for eligibility. Population: For 1 participant in Part 2, ECOG Performance was not given.
  Participants
    0 Fully active, able to carry on all pre-disease | 4 | 5 | 5 | 4 | 4 | 18 | 13 | 53
    1 Restricted in physically strenuous activity but ambulatory and able to carry out work | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 5
Pre-Treatment Tumor Size [Mean (Standard Deviation); unit: centimeters] — Length of longest diameter of tumor measured in centimeters. Population: For 1 participant in Part 3, pre-treatment tumor size was not reported.
  centimeters
    number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 19 | 13 | 57
    (all) | 2.9 (.84) | 4.06 (1.44) | 4.82 (2.03) | 3.76 (2.56) | 1.96 (0.82) | 4.13 (2.67) | 5.43 (2.19) | 4.03 (2.38)
American Joint Committee on Cancer (AJCC) Tumor Staging [Count of Participants; unit: Participants] — Participants had their tumors surgically removed and pathologically staged using the AJCC Staging criteria.
  Stage 1 breast cancer means that the cancer is small and only in the breast tissue or it might be found in lymph nodes close to the breast.
  Stage 2 breast cancer means that the cancer is either in the breast or in the nearby lymph nodes or both.
  Stage 3 means that the cancer has spread from the breast to the lymph nodes close to the breast, to the skin of the breast or to the chest wall.
  Stage 4 breast cancer has spread to another part of the body. Population: For 2 participants, both in Part 2, AJCC stage was not given.
  Participants
    number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 18 | 14 | 57
    Stage IA | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 4
    Stage IB | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
    Stage II | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 5
    Stage IIA | 1 | 2 | 0 | 1 | 1 | 4 | 2 | 11
    Stage IIB | 3 | 1 | 2 | 1 | 2 | 4 | 4 | 17
    Stage III | 0 | 0 | 0 | 1 | 0 | 3 | 2 | 6
    Stage IIIA | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 4
    Stage IIIB | 1 | 1 | 2 | 0 | 1 | 2 | 1 | 8
    Stage not reported/given | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Tumor Grade [Count of Participants; unit: Participants] — Participants had their tumors surgically removed and based off microscopic appearance of abnormality in cells, tumor was pathologically graded with the classifications Grade 1 (or well differentiated) means the cells are slower-growing, and look more like normal breast cells.
  Grade 2 (or moderately differentiated) means the cells are growing at a speed of and look like cells somewhere between grades 1 and 3.
  Grade 3 (poorly differentiated) means the cancer cells look very different from normal cells and will probably grow and spread faster.
  Grad X means the cancer cells cannot be assessed.
  Participants
    Grade I | 0 | 0 | 1 | 0 | 0 | 2 | 3 | 6
    Grade II | 2 | 4 | 2 | 3 | 2 | 9 | 4 | 26
    Grade III | 3 | 1 | 2 | 2 | 3 | 8 | 6 | 25
    Grade X (Unknown) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Tumor Type [Count of Participants; unit: Participants] — Luminal A or B tumor type
  Participants
    Luminal A | 2 | 4 | 3 | 2 | 1 | 0 | 0 | 12
    Luminal B | 3 | 1 | 2 | 3 | 4 | 0 | 0 | 13
    Not collected | 0 | 0 | 0 | 0 | 0 | 19 | 14 | 33

OUTCOME MEASURES:

1. Primary Outcome: Identify a Feasible Schedule of Vaccination Relative to SoC Neoadjuvant Chemotherapy When the Chemovax Are Administered Concurrently.
Description: Number of participants with sufficiently high anti-P10s immunoglobulin-G response Feasibility will be evaluated in terms of
  1. Generation of a sufficiently high anti-P10s immunoglobulin-G response
  2. Safety and tolerability of the combination of vaccine and chemotherapy
Time Frame: At the time of definitive surgery (4-8 weeks after chemo, which is between Week 22 and Week 25)
Population: This was defined as a >4-fold increase in a subject's anti-P10s-MAP IgG titer at Week 7 or later (at least 4 weeks after the 3rd immunization) relative to her pre-immune titer. For 1 participant, the Week 7 antibody titer was NA.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 - Chemovax Schedule A | Part 1 - Chemovax Schedule B | Part 1 - Chemovax Schedule C | Part 1 - Chemovax Schedule D | Part 1 - Chemovax Schedule E
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5
Participants
  Greater than or equal to 4-fold increase | 3 | 2 | 4 | 2 | 4
  Less than 4-fold increase | 2 | 3 | 1 | 3 | 1

2. Primary Outcome: Determine the pCR Rate
Description: The patient-level primary outcome for this objective is pathological Complete Response (pCR), which is binary yes/no, and the study-level endpoint for this outcome is the rate of pCR, i.e. the percentage of patients that achieved pCR=yes. The patient is assessed at the time of surgery for whether they achieved pCR=yes. They have to do the surgery in order to obtain the tissue samples on which they do their pCR assessment. Pathological Complete Response is defined as the absence of any residual invasive cancer on hematoxylin and eosin evaluation of the resected breast specimen and all sampled ipsilateral lymph nodes following completion of neoadjuvant systemic therapy (i.e., ypT0N0 or ypTisN0 in the AJCC staging system for staging solid tumors in the neoadjuvant setting that was described in a 2014 FDA Guidance for Industry).
Time Frame: At the time of definitive surgery (4-8 weeks after chemo, which is between Week 22 and Week 25)
Population: Clinical Response was determined for participants in Part 2 and 3. Part 2 Chemovax Schedule C was Stage 1 of the Simon 2-stage design. Stage 1's efficacy decision was a rule-based decision. If Stage 1 had 2 or more pCRs, then we could open up Stage 2 and start enrolling patients on it. Part 3 Chemovax Schedule C was Stage 2 of the Simon 2-stage design. It was supposed to enroll 22 subjects, but it had enrolled only 14 subjects by the time the study was closed to enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 - Chemovax Schedule A | Part 1 - Chemovax Schedule B | Part 1 - Chemovax Schedule C | Part 1 - Chemovax Schedule D | Part 1 - Chemovax Schedule E | Part 2 - Chemovax Schedule C | Part 3 - Chemovax Schedule C
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 19 | 14
Participants | 0 | 0 | 0 | 0 | 0 | 3 | 1

3. Secondary Outcome: P10s-MAP-Reactive Immunoglobulin Titers
Description: The anti-P10s binding level was measured via ELISA method after incubation with a subject's serum or plasma sample. Data was collected at multiple timepoints throughout the study. Values were averaged for each group.
Time Frame: Week 1 through Week 70
Measure: Mean (Standard Deviation); unit: titers
Arm/Group | Part 1 - Chemovax Schedule A | Part 1 - Chemovax Schedule B | Part 1 - Chemovax Schedule C | Part 1 - Chemovax Schedule D | Part 1 - Chemovax Schedule E
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5
titers | 10.72 (14.97) | 9.76 (13.91) | 42.25 (71.94) | 4.38 (5.10) | 6.74 (7)

4. Secondary Outcome: Activation Profiles of NK Cells: Pre-Immune and Post-Immune CD16
Description: Activated-NK-cell profiles will be determined via flow cytometry as the expression levels of different activation markers on NK cells in the subject's blood sample. Data was collected at multiple timepoints throughout the study. Values were averaged for each group. For some participants, CD16 was not assessable.
Time Frame: Week 1 through Week 70
Measure: Mean (Standard Deviation); unit: Median Fluorescence Intensity (MFI)
Arm/Group | Part 1 - Chemovax Schedule A | Part 1 - Chemovax Schedule B | Part 1 - Chemovax Schedule C | Part 1 - Chemovax Schedule D | Part 1 - Chemovax Schedule E | Part 2 - Chemovax Schedule C | Part 3 - Chemovax Schedule C
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 4 | 19 | 14
Median Fluorescence Intensity (MFI)
  Pre-Immune CD16 | 26065 (7976.46) | 26580 (2261.51) | 25171.8 (6493) | 28546 (7197.16) | 24897 (5334.72) | 67445.83 (31389.28) | 68619.59 (27944.66)
  Post-Immune CD16 | 19745.4 (5182.72) | 20993.4 (7061.48) | 27998.6 (10142.41) | 22959.8 (6020.06) | 25711.75 (20572.69) | 62323.05 (24021.75) | 65410.12 (24645.52)

5. Secondary Outcome: Activation Profiles of NK Cells: Pre-Immune and Post-Immune CD69
Description: Activated-NK-cell profiles will be determined via flow cytometry as the expression levels of different activation markers on NK cells in the subject's blood sample. Data was collected at multiple timepoints throughout the study. Values were averaged for each group. For some participants, CD69 was not assessable.
Time Frame: Week 1 through Week 70
Measure: Mean (Standard Deviation); unit: Median Fluorescence Intensity (MFI)
Arm/Group | Part 1 - Chemovax Schedule A | Part 1 - Chemovax Schedule B | Part 1 - Chemovax Schedule C | Part 1 - Chemovax Schedule D | Part 1 - Chemovax Schedule E | Part 2 - Chemovax Schedule C | Part 3 - Chemovax Schedule C
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 4 | 19 | 14
Median Fluorescence Intensity (MFI)
  Pre-Immune CD69 | 268.2 (50.08) | 300.8 (88.02) | 291.4 (38.55) | 294.6 (57.27) | 296.25 (34.37) | 428 (133) | 445.5 (169.17)
  Post-Immune CD69 | 307 (72.29) | 329.6 (26.23) | 275 (25.25) | 278.4 (27.87) | 311.25 (16.76) | 489.44 (139.9) | 505.97 (161.11)

6. Secondary Outcome: Activation Profiles of NK Cells: Pre-Immune and Post-Immune NKp46
Description: Activated-NK-cell profiles will be determined via flow cytometry as the expression levels of different activation markers on NK cells in the subject's blood sample. Data was collected at multiple timepoints throughout the study. Values were averaged for each group. For some participants, NKp46 was not assessable.
Time Frame: Week 1 through Week 70
Measure: Mean (Standard Deviation); unit: Median Fluorescence Intensity (MFI)
Arm/Group | Part 1 - Chemovax Schedule A | Part 1 - Chemovax Schedule B | Part 1 - Chemovax Schedule C | Part 1 - Chemovax Schedule D | Part 1 - Chemovax Schedule E | Part 2 - Chemovax Schedule C | Part 3 - Chemovax Schedule C
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 4 | 19 | 14
Median Fluorescence Intensity (MFI)
  Pre-Immune NKp46 | 685.2 (390.469) | 590.4 (204.147) | 724.2 (422.436) | 794.2 (355.618) | 744.25 (251.998) | 1360.33 (638.97) | 1650.08 (878.64)
  Post-Immune NKp46 | 1391 (489.819) | 1115.6 (485.348) | 1084.2 (930.867) | 1168.2 (324.282) | 1505.5 (1031.69) | 1412.13 (645.68) | 1813.56 (879.38)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of consent through the duration of the study, which is approximately 16 months after the first vaccination.
Groups:
- Part 2 & 3 Combined - Chemovax Schedule C: Primary Efficacy - Chemovax Schedule C: Subjects will receive three weekly injections of P10s-PADRE/MONTANIDE™ ISA 51 VG vaccine (week 1,2,3), then first cycle of chemotherapy (week 4), and subsequent cycles of chemotherapy every 21 days (week 7,10,13,16,19,22,25).
  Chemovax - P10s-PADRE/ MONTANIDE™ ISA 51 VG + Doxorubicin + Cyclophosphamide + Docetaxel (or Paclitaxel): Eligible subjects will be enrolled and immunized by SC administration of P10s-PADRE vaccine on each of 3 separate occasions over a three-week period.
  The 33 subjects combined from Parts 2 and 3 had the exact same treatment (Schedule C). The final efficacy evaluation required us to combine the pCRs from both parts.
Arm/Group | Part 1 - Chemovax Schedule A | Part 1 - Chemovax Schedule B | Part 1 - Chemovax Schedule C | Part 1 - Chemovax Schedule D | Part 1 - Chemovax Schedule E | Part 2 & 3 Combined - Chemovax Schedule C
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 1/33
Serious Adverse Events (participants affected / at risk) | 4/5 | 4/5 | 3/5 | 1/5 | 3/5 | 19/33
Other Adverse Events (participants affected / at risk) | 5/5 | 5/5 | 5/5 | 5/5 | 5/5 | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 - Chemovax Schedule A (N=5) | Part 1 - Chemovax Schedule B (N=5) | Part 1 - Chemovax Schedule C (N=5) | Part 1 - Chemovax Schedule D (N=5) | Part 1 - Chemovax Schedule E (N=5) | Part 2 & 3 Combined - Chemovax Schedule C (N=33)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 6 (15)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Mucositis Oral (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vomitting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lung Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 5 (13)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (7)
White blood cell decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (9)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardia disorders - Other, specify (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Esophageal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GGT increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Investigations - Other, specify (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspareunia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 - Chemovax Schedule A (N=5) | Part 1 - Chemovax Schedule B (N=5) | Part 1 - Chemovax Schedule C (N=5) | Part 1 - Chemovax Schedule D (N=5) | Part 1 - Chemovax Schedule E (N=5) | Part 2 & 3 Combined - Chemovax Schedule C (N=33)
Anemia (Blood and lymphatic system disorders) | 1 (4) | 5 (27) | 5 (11) | 3 (10) | 1 (2) | 29 (144)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 4 (4)
Vertigo (Ear and labyrinth disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (6)
Blurred vision (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 6 (7)
Dry Eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (5)
Eye Pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Watering eyes (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 12 (13)
Abdominal distension (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 11 (17)
Constipation (Gastrointestinal disorders) | 2 (4) | 2 (2) | 1 (1) | 4 (6) | 2 (2) | 22 (34)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 3 (3) | 20 (30)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 13 (16)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (2) | 1 (3) | 2 (3) | 3 (4) | 3 (4) | 8 (14)
Hemorrhoids (Gastrointestinal disorders) | 3 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 3 (4) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 9 (15)
Nausea (Gastrointestinal disorders) | 3 (5) | 4 (6) | 4 (5) | 5 (8) | 4 (4) | 29 (72)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Vomitting (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (4) | 17 (29)
Chills (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 7 (7)
Edema limbs (General disorders) | 4 (7) | 2 (2) | 0 (0) | 2 (2) | 1 (2) | 9 (11)
Edema trunk (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Fatigue (General disorders) | 3 (7) | 3 (5) | 4 (5) | 4 (11) | 5 (19) | 30 (80)
Fever (General disorders) | 3 (3) | 3 (4) | 0 (0) | 2 (2) | 3 (5) | 6 (6)
General disorders and administration (General disorders) | 1 (1) | 0 (0) | 1 (2) | 2 (3) | 0 (0) | 9 (15)
Injection site reaction (General disorders) | 4 (8) | 5 (7) | 5 (9) | 5 (6) | 5 (8) | 30 (49)
Pain (General disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 15 (26)
Autoimmune disorder (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorectal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0) | 3 (6) | 2 (2) | 0 (0) | 12 (16)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Skin infection (Infections and infestations) | 1 (3) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 3 (4)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 7 (8)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 3 (3)
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 6 (8)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 9 (15)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 15 (21)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 10 (17)
Creatinine increased (Investigations) | 1 (1) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 5 (20)
GGT increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 6 (9)
Investigations - Other, specify (Investigations) | 0 (0) | 4 (7) | 4 (6) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (3) | 5 (13) | 4 (11) | 1 (3) | 0 (0) | 26 (121)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 3 (13) | 5 (8) | 3 (7) | 18 (36)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 2 (4) | 2 (2) | 1 (1) | 8 (20)
Weight gain (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
White blood cell decreased (Investigations) | 1 (2) | 1 (2) | 3 (4) | 1 (2) | 1 (1) | 13 (35)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 2 (2) | 3 (4) | 3 (3) | 16 (23)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (7)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 13 (26)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 13 (42)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 16 (48)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 10 (23)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 11 (17)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (5) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 17 (25)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (5) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 6 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 14 (21)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 6 (11)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 13 (21)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 14 (20)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 3 (3) | 1 (1) | 2 (6) | 18 (23)
Dizziness (Nervous system disorders) | 1 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 15 (20)
Dysgeusia (Nervous system disorders) | 2 (2) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 6 (7)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 3 (9) | 0 (0) | 3 (3) | 3 (4) | 22 (42)
Memory impairment (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (5) | 1 (2) | 4 (4)
Parethesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 10 (13)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 3 (4) | 1 (1) | 1 (3) | 1 (1) | 10 (11)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus pain (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 19 (31)
Depression (Psychiatric disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 12 (17)
Insomnia (Psychiatric disorders) | 1 (2) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 18 (30)
Personality change (Psychiatric disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 7 (8)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (5)
Renal calculi (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 9 (19)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Reproductive system and breast disorder - Other, specify (Reproductive system and breast disorders) | 1 (3) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 7 (10)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (2) | 2 (3) | 0 | 1 (1) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 12 (16)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 11 (15)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 5 (8)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 6 (8)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 8 (10)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (6) | 0 (0) | 2 (2) | 2 (2) | 19 (24)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Erythema multifore (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 6 (6)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 6 (6)
Nail loss (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 3 (3)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (10)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 7 (7)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 3 (4) | 3 (4) | 1 (1) | 22 (39)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (5)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Hematoma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 1 (3) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 16 (20)
Hypertension (Vascular disorders) | 1 (2) | 3 (4) | 2 (6) | 0 (0) | 1 (1) | 12 (18)
Lymphedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 4 (4)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (7)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endocrine disorders - Other, specify (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flashing lights (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Optic nerve disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (12)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral dysesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Salivary duct inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Edema face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (10)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (12)
Cholesterol high (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INR increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Investigations - Other, specify (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 25 (143)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Metabolisms and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 11 (17)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (12)
dysesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spasticity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysmenorrhea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Irregular menstruatino (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Premature menopause (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Vaginal dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal hemorrhgae (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Body odor (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Scalp pain (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Social circumstances - Other, specify (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-02): https://cdn.clinicaltrials.gov/large-docs/84/NCT02229084/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/84/NCT02229084/ICF_002.pdf